CLINICAL TRIAL: NCT01343498
Title: A Phase I PK/PD Study of the PI3 Kinase/mTOR Inhibitor BEZ235 Given Twice Daily for the Treatment of Patients With Advanced Solid Tumors
Brief Title: Study of PI3 Kinase/mTOR Inhibitor BEZ235 Twice Daily for Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI REFMAL 233
Record Dates: First submitted 2011-04-22; First posted 2011-04-28 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Malignant Solid Tumour
Keywords: Solid Tumor Malignancy; Advanced Solid Tumors; BEZ235; mTOR Inhibitor
MeSH Terms: interventions — dactolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BEZ235 (Experimental)
  Interventions: Drug: BEZ235

INTERVENTIONS:
Drug: BEZ235 — BEZ235 will be given on a dose-escalation design, beginning at 200 mg BID (SDS sachet) in 3 patients and progressing to 400 mg, 600 mg, and 800 mg respectively based on tolerability.

SUMMARY:
This is a dose escalation trial to evaluate twice daily dosing of the sachet formulation of BEZ235. This trial will find the maximum tolerated dose (MTD) of the sachet formulation given twice daily, as well as evaluate pharmacokinetics (PK) and pharmacodynamics (PD) of the twice daily dosing. Patients will initially be given once daily dosing to determine the PK and PD of the single daily dose. On Day 9, they will begin twice daily dosing, with half of the single daily dose divided twice daily, and PK and PD of the twice daily dose will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of solid tumor malignancy that is metastatic or unresectable and not responsive to standard therapies or for which there is no effective therapy.
2. Eastern Cooperative Group (ECOG) Performance Status score of 0 or 1.
3. Patient has recovered (to grade ≤ 1) from all clinically significant toxicities related to prior antineoplastic therapies with the exception of alopecia and bone marrow and organ functions (described separately).
4. Adequate organ system function, defined as follows:

   • Absolute neutrophil count (ANC) ≥ 1.5 x 109/L

   • Platelets ≥ 100 x 109/L
   * Hemoglobin ≥ 9 g/dL
   * INR ≤ 2
   * Fasting plasma glucose ≤ 140 mg/dL
   * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 x the upper limit of normal (ULN) if no liver involvement or ≤ 5 x the upper limit of normal with liver involvement.
   * Creatinine ≤ 1.5 x ULN, OR calculated creatinine clearance ≥ 50 mL/min as calculated by the Cockcroft-Gault method, OR 24-hour measured urine creatinine clearance ≥ 50 mL/min.
5. Ability to swallow and retain oral medication.
6. Life expectancy of ≥ 3 months.
7. Male patients willing to use adequate contraceptive measures.
8. Female patients who are not of child-bearing potential, and female patients of child-bearing potential who agree to use adequate contraceptive measures and who have a negative serum or urine pregnancy test within 72 hours prior to initial trial treatment.
9. Patients must have measurable or evaluable disease.
10. Patients must be ≥18 years of age.
11. Patients entering this study must be willing to provide tissue from a previous tumor biopsy (if available) for correlative testing. If tissue is not available, a patient will still be eligible for enrollment into the study.
12. Ability to understand the nature of this trial and give written informed consent.

Exclusion Criteria:

1. Patients currently receiving cancer therapy (i.e., chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy [with the exception of LHRH agonists for prostate cancer], surgery and/or tumor embolization).
2. Use of an investigational drug within 21 days or 5 half-lives (whichever is shorter) prior to the first dose of BEZ235. For investigational drugs for which 5 half-lives is less than 21 days, a minimum of 10 days between termination of the investigational drug and administration of BEZ235 is required. In addition, any drug-related toxicity should have recovered to grade 1 or less.
3. Any major surgery, radiotherapy, or immunotherapy within the last 28 days (limited palliative radiation is allowed ≥ 2 weeks). Chemotherapy regimens with delayed toxicity within the last 4 weeks (or within the last 6 weeks for prior nitrosourea or mitomycin C). Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within the last 2 weeks.
4. Patient has received wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) ≤ 28 days or limited field radiation for palliation ≤ 14 days prior to starting study drug or has not recovered from side effects of such therapy.
5. Leptomeningeal metastases or spinal cord compression due to disease.
6. Patients with previously untreated brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if there is no evidence of central nervous system (CNS) disease progression, and at least 2 weeks have elapsed since treatment. Patients are not permitted to receive enzyme inducing anti-epileptic drugs (EIAEDs) during the study and should not be receiving chronic corticosteroid therapy for CNS metastases.
7. Patients with acute or chronic pancreatitis.
8. Patients with diabetes mellitus requiring insulin treatment or a history of gestational diabetes mellitus.
9. Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of BEZ235 (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea ≥ grade 2, and malabsorption syndrome).
10. Patient has active cardiac disease including any of the following:

    • Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)

    • QTcF > 480 msec on screening ECG
    * Unstable angina pectoris
    * Ventricular arrhythmias except for benign premature ventricular contractions
    * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
    * Conduction abnormality requiring a pacemaker
    * Valvular disease with documented compromise in cardiac function
    * Symptomatic pericarditis
11. Patient has a history of cardiac dysfunction including any of the following:

    * Myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV).
    * Documented cardiomyopathy
12. Family history of congenital long or short QT, or known history of QT/QTc prolongation or Torsades de Pointes (TdP). Patients who are currently receiving treatment with medication that has the potential to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug.
13. Inadequately controlled hypertension (i.e., SBP > 180 mmHg or DBP>100mmHg).
14. Patient is receiving chronic treatment with systemic steroids or another immuno-suppressive agent at the start of study treatment.

    Note: Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops, or local injections (e.g. intra-articular) are allowed.
15. Patient is consuming Seville oranges, grapefruit, grapefruit hybrids, pummelos or exotic citrus fruits (as well as their juices) during the last 7 days prior to start of treatment. Regular orange juice is permitted.
16. Patients who are receiving a strong CYP3A4 inhibitor or inducer.
17. Patients who are currently receiving treatment with therapeutic doses of warfarin sodium. Patients receiving low molecular weight heparin are allowed.
18. A serious active infection at the time of treatment, or another serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
19. Known diagnosis of human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C.
20. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
21. Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol.
22. Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol.
23. Women of child-bearing potential who are pregnant or breastfeeding or adults of reproductive potential not employing an effective method of birth control.

    * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 20 pg/mL] or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
    * Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the study and for 5 T1/2 (8 days) after stopping treatment. The highly effective contraception is defined as either:

1. True abstinence: When this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

2. Sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.

3. Male partner sterilization: (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female subjects on the study, the vasectomised male partner should be the sole partner for that patient.

4. Use of a combination of any two of the following (a+b):

1. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
2. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

Oral contraception, injected or implanted hormonal methods are not allowed as BEZ235 potentially decreases the effectiveness of hormonal contraceptives.

* Women of child-bearing potential must have a negative serum or urine pregnancy test ≤ 72 hours prior to initiating treatment.
* Fertile males, defined as all males physiologically capable of conceiving offspring must use condom during treatment, for 5 T1/2 (8 days) after stopping treatment and for additional 12 weeks (3 months in total after study drug discontinuation) and should not father a child in this period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of BEZ235 given twice daily | 18 months
  To determine the maximum tolerated dose (MTD) of BEZ235 given twice daily in patients with advanced solid tumors

SECONDARY OUTCOMES:
To describe the toxicities of this regimen | 18 months
  The safety endpoints to be summarized are:
  * Incidence of dose-limiting toxicities (DLTs)
  * Incidence of adverse events (AEs)
  * Incidence of grade 1, grade 2, grade 3 and grade 4 AEs
  * Incidence of serious adverse events (SAEs)
Clinical Efficacy | 18 months
  To describe the clinical efficacy of this regimen in patients with advanced solid tumors. The tumor response will be measured by the number of patients with complete responses, partial responses, stable disease and progressive disease.
PK profile of BEZ235 | 18 months
  To characterize the PK profile of BEZ235 given as a twice daily dose. The PK parameters (including AUC (0-∞), AUC (0-t), Cmax, tmax, λz, and t½) of BEZ235 following oral administration will be assessed by analysis of BEZ235 plasma concentrations using a non-compartmental approach.
  During treatment PK blood samples will be taken at the following timepoints:
  * Cycle 1, Day 1: pre-dose, 1, 2, 4, 8, 10, 12 and 24 hours post-dose
  * Cycle 1, Day 8: pre-dose, 1, 2, 4, 8, 10, 12 and 24 hours post-dose
  * Cycle 1, Day 28: pre-dose, and at 1, 2, 4, 8, 10, 12 and 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Johanna C Bendell, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (2):
- United States (2):
  - Oklahoma University, Oklahoma City, Oklahoma
  - Tennessee Oncology, Nashville, Tennessee